CLINICAL TRIAL: NCT01726439
Title: A 5-year Prospective and Observational Study to Evaluate the Effectiveness of Nucleos(t)Ide Analogs (NUC) Therapy Among Chronic Hepatitis B (CHB) Patients Naive to NUC in Real World Practice at Hospitals in Tier 2 Cities in China (the EVOLVE Study)
Brief Title: Effectiveness of Nucleos(t)Ide Analogs (NUC) Therapy Among Naive CHB Patients in China
Acronym: EVOLVE
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: AI463-952
Record Dates: First submitted 2012-11-06; First posted 2012-11-15 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CHB patients who are naive to NUC treatment: CHB patients who are naive to NUC at enrollment and be treated at hospitals at tier 2 cities in China

SUMMARY:
To compare the effectiveness, in a real world practice setting in tier 2 cities of China, of Entecavir (ETV) monotherapy and Lamivudine (LAM) based therapies (including LAM monotherapy, de novo LAM + Adefovir [ADV] combination, and early add-on of ADV) among chronic hepatitis B (CHB) patients who are naive to NUC at enrollment to this study

DETAILED DESCRIPTION:
Sampling Method: Consecutive patient sampling

Biospecimen Retention: Blood samples for HBV viral load testing along the treatment period of this study

ELIGIBILITY:
Inclusion Criteria:

* CHB patients, or CHB patients with compensated cirrhosis, as defined by the current Chinese guidelines
* Male or female
* ≥ 18 years of age
* Either Hepatitis B e antigen (HBeAg) positive or negative
* Naïve to NUC (defined as no previous exposure to NUC treatment as based on patient self-report)
* Has compensated liver disease
* Patients with compensated cirrhosis
* Patients who consent to participate in this study
* Local residents with medical reimbursement coverage preferred

Exclusion Criteria:

* Co-infected with hepatitis C virus (HCV)
* CHB patients with decompensated cirrhosis, liver failure, hepatocellular carcinoma, or any other types of malignancy at the screening phase
* CHB patients who are being treated by interferon therapy within 6 months immediately prior to the screening phase of this study
* CHB patients with a confirmed pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals in Chinese tier 2 cities. The definition of these hospitals is the following:
  * Hospitals where 300 or more CHB patients are treated monthly
  * Hospitals where PCR can be performed in the hospital's laboratory to measure HBV DNA serum levels
Sampling Method: Non-Probability Sample
Enrollment: 3434 (Actual)
Dates: Start 2012-12; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve virology response (defined as HBV DNA < 300 copies/mL) by ETV monotherapy in comparison with LAM-based therapy | 48 weeks after initial NUC antiviral therapy
  Virology response is defined as Hepatitis B virus (HBV) Deoxyribonucleic acid (DNA) < 300 copies/mL by a highly sensitive assay such as Roche COBAS or Abbott Real Time Polymerase chain reaction (PCR) performed in a one central laboratory

SECONDARY OUTCOMES:
Mean HBV DNA reductions after 48 weeks of treatment from baseline for ETV and LAM-based therapy patients (stratifying by the 3 LAM-based subgroups) | Baseline (Day 1) and 48 weeks
Proportion of patients who achieve virology response by ETV in comparison with LAM-based therapy after 24 weeks and 96 weeks of treatment (stratifying by the 3 LAM based subgroups) | 24 weeks and 96 weeks
Proportion of patients who modify their initial treatment options to manage suboptimal response or resistance after 24 weeks, 48 weeks, and 96 weeks of treatment among all treatment options | 24 weeks, 48 weeks and 96 weeks
Proportion of patients who achieve virology response among other treatment options, including ADV, LdT, and combinations of NUCs, after 24 weeks, 48 weeks, 72 weeks, 96 weeks, 144 weeks, 192 weeks and 240 weeks of treatment | 24 weeks, 48 weeks, 72 weeks, 96 weeks, 144 weeks, 192 weeks and 240 weeks
  HBV DNA levels at week 24 will be analyzed at the laboratories of hospitals where the patients are treated while evaluation of HBV DNA levels after 48 and 96 weeks of treatment will be conducted at the central laboratory
Cumulative incidence of patients who develop viral breakthrough and/or genotypic resistance | 24 weeks, 48 weeks, 72 weeks, 96 weeks, 144 weeks, 192 weeks and 240 weeks
Cumulative incidence of clinical outcome (eg, HCC, death, decompensated cirrhosis) in ETV arm versus LAM-based and other treatment arms | 48 weeks, 96 weeks, 144 weeks, 192 weeks and 240 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (44):
- China (44):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Fuzhou, Fujian
  - Local Institution, Quanzhou, Fujian
  - Local Institution, Xiamen, Fujian
  - Local Institution, Foshan, Guangdong
  - Local Institution, Shenzhen, Guangdong
  - Local Institution, Nanning, Guangxi
  - Local institution, Guiyang, Guizhou
  - Local Institution, Guiyang, Guizhou
  - Local Institution, Haikou, Hainan
  - Local Institution, Baoding, Hebei
  - Local Institution, Shijiazhuang, Hebei
  - Local Institution, Daqing, Heilongjiang
  - Local Institution, Haerbin, Heilongjiang
  - Local Institution, Zhengzhou, Henan
  - Local Institution, Shiyan, Hubei
  - Local Institution, Wuhan, Hubei
  - Local Institution, Changsha, Hunan
  - Local Institution, Ordos, Inner Mongolia
  - Local Institution, Changshu, Jiangsu
  - Local Institution, Changzhou, Jiangsu
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Nangchang, Jiangxi
  - Local Institution, Changchun, Jilin
  - Local institution, Yanji, Jilin
  - Local Institution, Dalian, Liaoning
  - Local Instution, Fushun, Liaoning
  - Local Institution, Shengyang, Liaoning
  - Local Institution, Shenyang, Liaoning
  - Local Institution, Yinchuan, Ningxia
  - Local Institution, Jinan, Shandong
  - Local Institution, Qingdao, Shandong
  - Local Institution, Yantai, Shandong
  - Local Institution, Taiyuan, Shanxi
  - Local Institution, Xi’an, Shanxi
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Ürümqi, Xinjiang
  - Local institution, Hangzhou, Zhejiang
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Jinghua, Zhejiang
  - Local Institution, Ningbo, Zhejiang

REFERENCES:
- [Derived] Jia J, Shang J, Tang H, Jiang J, Ning Q, Dou X, Zhang S, Zhang M, Han T, Tan D, Zhou X, Chen G, Sheng J, Su Z, Chen H, Dai E, Ye Y, Guo Y, Shen Y, Yuan J, Wei Z, Zhu S; EVOLVE Study Group. Long-term outcomes in Chinese patients with chronic hepatitis B receiving nucleoside/nucleotide analogue therapy in real-world clinical practice: 5-year results from the EVOLVE study. Antivir Ther. 2020;25(6):293-304. doi: 10.3851/IMP3372. PMID 33090970
- [Derived] Jia J, Tang H, Ning Q, Jiang J, Dou X, Zhang M, Zhang S, Shang J, Lu W, Ye Y, Wang X, Li M, Liu J, Bo Q, Tan W; EVOLVE Study Group. Real-world evidence for nucleoside/nucleotide analogues in a 5-year multicentre study of antiviral-naive chronic hepatitis B patients in China: 52-week results. Antivir Ther. 2018;23(3):201-209. doi: 10.3851/IMP3205. PMID 29116050
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx